CLINICAL TRIAL: NCT03152383
Title: Examination of Differential Valuation of Leisure Items and Attention as Reinforcers in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nathan A. Call, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00056563; R21MH108873 (NIH)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Autism
Keywords: Autism Spectrum Disorder; Behavioral Research; Psychology; Cognitive Disorders
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Children with autism, typically developing children, and children with developmental disabilities will participate in the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autism Spectrum Disorder (Experimental): Children diagnosed as having autism spectrum disorder
  Interventions: Behavioral: Training trials; Behavioral: Progressive Ratio Session; Behavioral: Re-test; Behavioral: Pairing Protocol
- Typically developing (Active Comparator): Children who are typically developing
  Interventions: Behavioral: Training trials; Behavioral: Progressive Ratio Session
- Other Developmental Delay (Active Comparator): Children diagnosed with a developmental delay other than autism spectrum disorder
  Interventions: Behavioral: Training trials; Behavioral: Progressive Ratio Session

INTERVENTIONS:
Behavioral: Training trials — A highly preferred edible item will be selected to teach the contingencies for the assessment. Materials to engage in the work response (i.e., button press) will be placed within arm's reach of the child, and the edible item will be in sight. The therapist will deliver a vocal prompt for the child to engage in the work response (e.g., "press the button and you can have some candy"). If the child engages in the response, the therapist immediately delivers the edible item. The therapist will guide the child to engage in the instrumental response, and will then gradually begin to fade the prompt level. If the child makes an error at any level of prompting, the therapist will guide the participant to emit a correct response. The edible item will be delivered to the child each time that the child responds correctly at any prompt level.
Behavioral: Progressive Ratio Session — The child will be guided to engage in the instrumental response then the stimulus will be immediately delivered for 30 seconds. The leisure item or the individual who will provide attention will be directly outside of the session room. If the child emits the work response, they will be allowed access to either a leisure item or to attention (depending on the condition) for 30 seconds. The child is initially required to respond one time, then they will be required to respond two times to gain access to the item or attention (then 4, then 8, and so on) such that the response requirement progressively increases according to a pre-determined schedule. A minimum of 3 sessions will be conducted for each condition. The amount of time required for participation depends on the child's responding, and caregiver availability. Participation may take as little as a couple hours, or as long as 3-4 hours per day for approximately one week.
Behavioral: Re-test — 10 children with ASD will return to repeat the progressive ratio (PR) assessment one week after completing it the first time to examine the reliability of the measure.
  Arms: Autism Spectrum Disorder
Behavioral: Pairing Protocol — 15 children with ASD will receive an intervention designed to increase social approach after completing the PR assessment. Participants will attend 2 hour appointments 3-5 days per week in which a therapist will deliver highly preferred items, play with the child, work on teaching communication skills, and teach the child to comply with demands. After completing the intervention (once the child is willingly staying near and interacting with the therapist and complying with instructions), the PR assessment will be repeated to measure change due to the intervention.
  Arms: Autism Spectrum Disorder

SUMMARY:
The purpose of this study is to compare how children with autism, typically developing children, and children with other developmental delays value social attention and toys. The first part of the study seeks to determine whether breakpoints when responding on progressive ratio (PR) schedules can be used to determine the value of leisure items and attention. By comparing the breakpoints obtained for leisure items and attention, the researchers will determine the differential valuation of leisure items and attention. It is anticipated that the manner in which individuals with an autism spectrum disorder (ASD) diagnosis and those who do not will differ with respect to the degree to which they value these two types of stimuli. The second part of the study seeks to determine whether an intervention in which social attention is paired with primary reinforcers impacts responding during the PR assessment, in children with ASD.

DETAILED DESCRIPTION:
The three core features of autism spectrum disorder (ASD) are impairments in social interaction, restricted range of interest, and stereotyped/repetitive behavior. However, autism is a heterogeneous disorder, and individuals with a diagnosis vary widely in specific presentation. For example, despite an overall impairment in social behavior, some individuals with an autism diagnosis still frequently initiate social interactions with others. In contrast, others may engage in problem behaviors maintained by escape or avoidance of social interactions.

A progressive ratio (PR) assessment is one method for directly quantifying the degree to which an individual values a particular stimulus or event. Within a PR assessment, reinforcement occurs under schedule requirements that increase following each set of responses within a single session until responding ceases. The highest schedule requirement completed (i.e., breakpoint) can then be used as a measure of how much an individual is willing to respond for a given stimulus.

The study will include about 65 children, 25 children with ASD and 15 typically developing children, and 25 children with developmental disabilities other than ASD. Children with autism, typically developing children, and children with non-ASD developmental delays other than ASD will be compared in terms of how they value social attention and toys. The child participants will be asked to do an action, such as pressing a button, to receive either an item or attention. At first, the participants will only be required to do the action once, but after the first time the children will be required do more and more before they can get the item or attention. Eventually, most children stop responding for the preferred item or attention. The study will consider the child as done working when they go for one minute without performing the action. Sessions will end after 30 minutes if the child keeps working without stopping. This study will examine how many times the child will respond for items and attention. 15 of the children with ASD will be asked to come back for an additional appointment one week after they complete the assessment of how they value attention and toys. The PR assessment will be repeated see if the children respond the same way at different times.

The second part of the study will include 10 children diagnosed with ASD ranging in age from two to six. All of the procedures described in part one of the study will be included. The PR assessment will be completed prior to intervention and again after intervention. All appointments will be conducted over a maximum of 4 weeks. The intervention will be based on the principals of respondent conditioning; social interaction will be paired with the delivery of other reinforcers, such as edible items, to increase the value of social interaction. Sessions will be conducted 5 days per week and will be up to two hours long. Following the intervention, the participant will repeat the PR assessment in order to assess whether the intervention increased the value of social interaction.

ELIGIBILITY:
Inclusion Criteria for Autism Spectrum Disorder (ASD) Group:

* Between the ages of 3 and 6.
* Presence of an autism diagnosis as determined by The Autism Diagnostic Observation Schedule (ADOS).
* Adaptive functioning typical of autism as determined by the Vineland Adaptive Behavior Scales (VABS-II; survey interview form).
* Completion of the Social Responsiveness Scale (SRS) to assess social impairment.
* Completion of the Early Social Communication Scales to assess non-verbal communication.

Inclusion Criteria for Typically Developing Group:

* Between the ages of 3 and 6.
* Current developmental level determined to be not developmentally delayed per The Mullen Scales of Early Learning (MSEL) or Differential Ability Scale (DAS; depending on participant age).

Inclusion Criteria for Other Developmental Delays Group:

* Between the ages of 3 and 6.
* Current developmental level determined to be developmentally delayed per The Mullen Scales of Early Learning (MSEL) or Differential Ability Scale (DAS; depending on participant age).

Exclusion Criteria for all groups:

* Caregiver does not give permission for protective procedures and emergency protocols to be used if the child participant exhibits problem behaviors during a study visit.
* Children who are not able to master the training trial within 10 sessions will not participate in the study.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2012-06-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Breakpoint achieved for each stimulus | Up to one week
  The highest schedule requirement completed (i.e., breakpoint) is used as a measure of how much an individual is willing to respond for a given stimulus.
Change in breakpoints | Assessment 1 through repeat assessment (up to 4 weeks)
  For children receiving the intervention the change between breakpoints across the two PR assessments conducted before and after intervention will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan A Call, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03152383/ICF_000.pdf